CLINICAL TRIAL: NCT06578884
Title: A Prospective Clinical Investigation to Evaluate the Safety and Performance of 877PTY Toric IOL for Visual Correction of Corneal Astigmatism
Status: Enrolling by invitation | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: M-877PTY-HU-2301
Record Dates: First submitted 2024-06-10; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Cataract; Corneal Astigmatism
Keywords: cataract; intraocular lens (IOL); astigmatism correction; aphakic
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 877PTY: 100 patients/eyes implanted with 877PTY IOL
  Interventions: Device: 877PTY

INTERVENTIONS:
Device: 877PTY — IOL implantation with 6-month follow-up period Monocular UDVA/CDVA Manifest Refraction (SPH, CYL, SEQ) Optical Biometry, Keratometry (K1, K2, AXL, ACD) IOL axis orientation determination Visual function questionnaire Glistening evaluation Tonometry Slit-Lamp examination Fundus visualization

SUMMARY:
Medicontur preloaded hydrophobic monofocal toric intraocular lenses (IOLs) are indicated to improve vision at far distance in adults with or without cataract and correction of pre-existing corneal astigmatism secondarily to removal of the crystalline lens.

The intraocular lens is intended to be surgically implanted into the eye with the purpose of restoring optical function in the aphakic eye to provide an optical system with high predictability of the precalculated dioptric power.

The investigation will be performed as a prospective, non-comparative, single arm study with a single center design. Patients will be enrolled who are assigned to be implanted with the 877PTY IOLs mono- or binocularly between January 2024 - June 2025.

Data from six visits will be collected:

* Visit 1: Screening and Baseline (up to 90 days prior to the surgery)
* Visit 2: IOL implantation (Day 0)
* Visit 3: Day 1 post-operatively (+/- 0 day)
* Visit 4: Day 7 post-operatively (+/- 3 days)
* Visit 5: Month 1 post-operatively (+/- 2 weeks)
* Visit 6: Month 6 post-operatively (+/- 1 month)

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years old and older);
* cataract and/or corneal astigmatism diagnosis;
* indication for cataract surgery or refractive lens exchange;
* recommended cylinder correction with toric IOL with cylinder power ≥1.0D;
* clear intraocular media other than cataract;
* signed informed consent form;

Exclusion Criteria:

* irregular astigmatism;
* patients who are not targeted to emmetropia (predicted residual spherical equivalent and/or astigmatism is out of the range of ±0.5D and ±0.38D respectively);
* any retinopathy or maculopathy that affects the vision;
* iris neovascularization;
* congenital eye abnormality affecting visual performance;
* advanced glaucoma;
* pseudoexfoliation syndrome affecting IOL stability;
* amblyopia;
* uveitis;
* retinal detachment;
* prior ocular surgery in personal medical history;
* irregular corneal curvature or corneal diseases affecting visual performance;
* high myopia (axial length ≥ 26,5 mm);
* inadequate visualization of the fundus on preoperative examination;
* dilated pupil size not large enough to visualize toric IOL axis markings postoperatively based on the Investigator's decision;
* eye trauma in medical history;
* instability of keratometry or biometry measurements;
* prior corneal refractive surgery such as LASIK, PRK, or SMILE;
* patients deemed ineligible by the investigator because of any systemic disease or treatment;
* pregnancy or lactation;
* current use of systemic steroids or external ophthalmic drugs;
* concurrent participation in another drug or device investigation.

Intraoperative exclusions: the presence of the following intraoperative exclusion criteria will lead to the exclusion of the subject:

- Any unexpected or serious intraoperative complication that makes IOL implantation impossible or results in implantation of another type of IOL that is outside the scope of this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aphakic adult patients (18 years old and older), with cataract and corneal astigmatism who aspire to have improved uncorrected distance vision and reduction of the residual refractive cylinder and assigned to monocular or binocular implantation with 877PTY IOL.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Performance Endpoint - CDVA | 6 months postoperatively
  Visual acuity: monocular CDVA at 6 months after IOL implantation

SECONDARY OUTCOMES:
Secondary Performance Endpoint - UDVA | 6 months postoperatively
  Visual acuity: monocular UDVA at 6 months after IOL implantation
Secondary Performance Endpoint - Subjective CYL | 6 months postoperatively
  Subjective (manifest) cylinder and keratometric cylinder of the eye at 6 months postoperatively
Secondary Performance Endpoint - Residual CYL and SEQ | 6 months postoperatively
  Residual manifest cylinder and spherical equivalent at 6 months postoperatively;
Secondary Performance Endpoint - Rotational stability | 6 months postoperatively
  IOL rotational stability at 6 months after IOL implantation;
Secondary Performance Endpoint - Injector handling | 6 months postoperatively
  Ease of IOL implantation and positioning at surgery;
Secondary Performance Endpoint - Patient satisfaction (VFQ-25) | 6 months postoperatively
  Patient-reported visual functions: overall global vision rating, difficulty with near and distance vision activities, social functioning and role limitations, dependency on others, mental health symptoms due to vision, driving difficulties, limitations with peripheral and color vision, and ocular pain evaluated by visual function questionnaire at 6 months after IOL implantation.
Secondary Performance Endpoint - Glistening | 6 months postoperatively
  Glistening rate and severity at 6 months after IOL implantation

OTHER OUTCOMES:
Safety Endpoints - Intraoperative complications | Up to day 1 postoperatively
  Intraoperative complications of cataract surgery
  * Posterior capsular or zonular rupture
  * Vitreous loss/anterior vitrectomy or aspiration
  * Iris/ciliary body injury
  * Loss of nuclear material into vitreous
  * Suprachoroidal haemorrhage
  * Retrobulbar haemorrhage
Safety Endpoints - Postoperative complications | Up to month 1 postoperatively
  Postoperative complications of cataract surgery
  * Cystoid macular oedema
  * Iris abnormalities
  * Corneal oedema
  * Wound leak or rupture
  * IOL dislocation, removal, or exchange
  * Inflammation (Endophthalmitis, anterior chamber cells, anterior chamber flare, hypopyon)
  * Retinal tear, break, or detachment
  * Persistent iritis
  * Elevated intraocular pressure
  * Pupillary block
  * Cornea status
Safety Endpoints - Complications of IOL implantation | Up to month 6 postoperatively
  Complications of IOL implantation
  * Posterior capsular opacification (PCO)
  * Opacification, IOL discoloration

CONTACTS AND LOCATIONS:
Locations (1):
- Győr-Moson-Sopron Vármegyei Petz Aladár Egyetemi Oktató Kórház, Győr, Hungary